CLINICAL TRIAL: NCT04523025
Title: Nordic Cystectomy Study I - Prospective Validation of Neutrophil/Lymphocyte Ratio as Predictor of Bladder Cancer Survival Risk After Radical Cystectomy for Bladder Cancer
Brief Title: Nordic Cystectomy Study I - Neutrophil-lymphocyte Ratio (NLR)
Acronym: NorCys-NLR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Nordic Urothelial Cancer Group (Other)
Responsible Party: Sponsor
Other Study IDs: T197/2020
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Bladder Cancer; Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low NLR-ratio: Patients with low NLR ratio (NLR<3)
  Interventions: Diagnostic Test: NLR-ratio
- High NLR-ratio: Patients with high NLR ratio (NLR≥3)
  Interventions: Diagnostic Test: NLR-ratio

INTERVENTIONS:
Diagnostic Test: NLR-ratio — The ratio of neutrophils and lymphocytes in patients blood sample prior to surgical operation

SUMMARY:
Around 7200 cases of Muscle Invasive Bladder Cancer are diagnosed annually in the Nordic countries combined. Muscle Invasive Bladder Cancer is an aggressive disease and it is linked with high mortality rates. The golden standard of treatment is radical cystectomy (RC) (the surgical removal of the bladder) and radical removal of lymph nodes in the pelvis. In addition to surgical treatment, and especially in cases where the tumour invades tissues surrounding the bladder or lymph nodes, chemotherapy is recommended. Chemotherapy can be administered before or after surgery, in a neoadjuvant (NAC) or adjuvant setting (AC). Although most patients recover well from surgery, there are significant risks regarding radical cystectomy. The greatest challenges in planning the treatment are making individual risk assessments and prognosis for the treated patients. Neoadjuvant chemotherapy is also insufficiently used and it is hard to predict how the tumour responds to chemotherapy.

The purpose of this study is to collect prospective clinical data on radical cystectomy -patients in co-operation with other Nordic countries: Sweden, Denmark, Iceland and Norway. The collected data is used to validate existing prediction tools and discover novel tools for prediction of morbidity related to RC and prediction of oncological outcome after RC. The study is divided into three sub-studies. The second sub-study is on the preoperative neutrophil-lymphocyte ratio (NLR). Some studies suggest that NLR might be a predictor of oncological outcome of BC after RC. In addition, NLR has been suggested to correlate with NAC response and outcome after NAC and RC. The used cut-off value for NLR has varied between 2.26-3.0.

Patients will be allocated into two groups: low NLR ratio (NLR<3), and high NLR ratio (NLR≥3). The lab test will be retrieved before RC at the time of routine clinical laboratory testing for all patients and also before the initiation of NAC for patients planned to have chemotherapy. The primary end-point is bladder-cancer specific survival and, and secondary endpoints include progression-free, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed urinary BC planned to be treated with RC with or without neoadjuvant chemotherapy.
2. Histologically confirmed urinary BC planned to be treated with palliative cystectomy 2) Signed informed consent 3) Patient age >18 years

Exclusion Criteria:

1. RC for other reasons than BC
2. Other forms of surgical treatment of BC than RC (e.g. bladder resection).
3. Patient unwillingness to participate in the study for any reason (i.e. lack of signed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with muscle-invasive bladder cancer undergoing radical cystectomy -surgery
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Bladder-cancer specific survival | 24 months

SECONDARY OUTCOMES:
Progression-free survival | 24 months
overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- University Hospital of Turku, Hospital Distric of Southwest Finland, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No